CLINICAL TRIAL: NCT07089238
Title: Exploring the Effects of Citicoline Supplementation on Validated Subjective and Objective Markers of Mood in Healthy Volunteers: A Randomized, Double-blind, Placebo-controlled, Parallel-group Trial
Brief Title: Evaluate the Effects of Citicoline on Mood in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirin Holdings Company, Limited (Industry)
Collaborators: The Center for Applied Health Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: KIRIN-01-2025
Record Dates: First submitted 2025-07-10; First posted 2025-07-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Cognitive; Citicoline; Cognitive performance; Mood
MeSH Terms: interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Intervention Model Description: There are 2 study groups, including one test product (TP) group and one placebo (PL) group. Healthy adult males and females who are 21 to 65 years of age (inclusive) at screening will be enrolled.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The placebo will match the TP in physical and visual appearance and packaging and each participant's study product assignments will be associated with a unique code to prevent premature unblinding. Planned unblinding will occur following database lock, definition of study populations, and a blinded statistical analysis. Delegated unblinded site personnel will be responsible for study product accountability, reconciliation, and record maintenance (i.e., receipt, reconciliation, and final disposition records) throughout the course of the study. The investigator will have oversight in a blinded manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citicoline (Active Comparator)
  Interventions: Dietary Supplement: Citicoline
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Citicoline — Oral
  Arms: Citicoline
Dietary Supplement: Placebo — Oral
  Arms: Placebo

SUMMARY:
The objective of this trial is to determine the effects of citicoline on mood in healthy Men and Women compared to a placebo.

DETAILED DESCRIPTION:
This study is a 4-week, randomized, double-blind, placebo-controlled trial of citicoline in healthy men and women. Cognitive assessments will be performed to determine whether citicoline administration improves mood, compared to placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health and able to participate as determined by medical history and routine blood chemistries.
* Biological men and women between 21 and 65 years of age (inclusive).
* Body Mass Index of 18.5-32.0 (inclusive).
* Body weight of at least 110 pounds.
* Participant is experiencing moderate levels of mood disturbance during screening.
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg.
* Normal supine, resting heart rate (<90 per minute).
* Agrees to maintain their existing dietary and physical activity patterns throughout the study period.
* Participants agree to maintain their usual caffeine consumption habits, given that they do not exceed the maximum intake per day (400mg/day or 3-4 cups of coffee per day).
* If a dietary supplement was initiated within the past month, the participant is willing to discontinue supplement use followed by a 2-week washout prior to participation in the study.
* Willing to duplicate their previous 24-hour diet, refrain from caffeine for 24 hours, refrain from alcohol and exercise for 24 hours prior to each trial, and fast for 10 hours prior to each visit.

Exclusion Criteria:

* QIDS (Quick Inventory of Depressive Symptomology) score > 16.
* Women who are pregnant, lactating, or planning to become pregnant during the study. Women must have a negative pregnancy test at screening.
* Women with a PSST (Premenstrual Symptoms Screening Tool) score ≥30
* Current smokers or cessation within 3 months prior to screening.
* Alcohol consumption (>2 standard alcoholic drinks/day or >10 drinks/week) or drug abuse/dependence.
* Current use of any nootropic dietary supplements (e.g., GABA, Ashwaghanda, St. John's Wort, Ginkgo biloba, L-theanine, choline, Lion's mane, creatine, etc.) or medications (e.g., piracetam, Adderall, modafinil, etc.) that may confound the study or its endpoints.
* Medical history of hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* Individuals who have been diagnosed with digestive, liver, renal, cardiovascular, or other metabolic diseases.
* Other known gastrointestinal or metabolic diseases that might impact nutrient absorption, distribution, metabolism, or excretion (e.g., intestinal malabsorption, electrolyte abnormalities, diabetes, thyroid disease, adrenal disease, hypogonadism, short bowel syndrome, diarrheal illnesses, history of colon resection, gastric ulcer, reflux disease, gastroparesis, Inborn-Errors-of-Metabolism, etc.).
* Chronic medically diagnosed inflammatory condition or disease (e.g., rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Medical history of a cognitive (i.e., ADD/ADHD) or psychiatric disorder, or brain-related medical conditions (e.g., TBI, ADHD).
* Currently using medications to treat anxiety or depression.
* Have an irregular sleep pattern (i.e. shift workers) or inadequate sleep schedule (i.e., less than 6 hours per night).
* Known sensitivity, allergy, or intolerability to any ingredient in the test products.
* Participants who report a clinically significant illness within the last 30 days.
* Individuals who are cognitively impaired and/or who are unable to give informed consent.
* Any other diseases or conditions that, in the opinion of the Principal Investigator, could confound the primary endpoint or place the subject at increased risk of harm if they were to participate.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Total Mood Disturbance (TMD) score on the Profile of Mood States second eddition-Adult short (POMS2) | 4 weeks
  To evaluate the effect of the Test Product (TP) on TMD on the POMS2 compared to a placebo

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 4 weeks
  To evaluate the effect of the TP on PSQI compared to a placebo
Perceived Stress Scale (PSS-10) | 4 weeks
  To evaluate the effect of the TP on PSS-10 compared to a placebo
Serum Brain-Derived Neurotrophic Factor (BDNF) and Homovanilic Acid (HVA) | 4 weeks
  To evaluate the effect of the TP on serum BDNF and HVA compared to a placebo
Profile of Mood States second eddition-Adult short (POMS2) subdomain scores | 4 weeks
  To evaluate the effect of the TP on POMS2 subdomain scores compared to a placebo

OTHER OUTCOMES:
Adverse events | 0-4 weeks
  To assess the safety and tolerability of the TP in healthy participants: Reports of Adverse Events to determine number of participants with adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States